CLINICAL TRIAL: NCT04876768
Title: Effects of High Intra-procedural Oxygen Fraction on Post-ERCP Pancreatitis: A Randomized Clinical Trial
Brief Title: Effects of High FIO2 on Post-ERCP Pancreatitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syed Z. Ali, MD (Other)
Responsible Party: Sponsor-Investigator, Syed Z. Ali, MD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 56565
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Post-ERCP Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Endoscopist will be blinded but the anesthetist will not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of 80% oxygen(high oxygen fraction) during ERCP (Experimental): Anesthetist will open the envelope of randomly assigned groups which will assign patients to 80% FIO2(supplemental perioperative high oxygen fraction). 80% FIO2 will be maintained during the ERCP procedure. Maintaining oxygen saturation of > 92% through administration of oxygen via nasal cannula, mask or ventilator will be per anesthetist discretion. Additional supplemental oxygen will be given to patients at any time, as necessary, to maintain oxygen saturation as measured by pulse oximeter > 92%.
  Interventions: Procedure: Use of different concentrations of oxygen during ERCP
- Use of 30% oxygen(normal oxygen fraction) during ERCP (Active Comparator): Anesthetist will open the envelope of randomly assigned groups which will assign patients to 30% FIO2 (normal oxygen fraction). 30% FIO2 will be maintained during the ERCP procedure. Maintaining oxygen saturation of > 92% through administration of oxygen via nasal cannula, mask or ventilator will be per anesthetist discretion. Additional supplemental oxygen will be given to patients at any time, as necessary, to maintain oxygen saturation as measured by pulse oximeter > 92%.
  Interventions: Procedure: Use of different concentrations of oxygen during ERCP

INTERVENTIONS:
Procedure: Use of different concentrations of oxygen during ERCP — The endoscopic intervention will be conducted in the endoscopy suite located at UK Albert B. Chandler Hospital in Lexington, Kentucky. ERCP/EUS uses an endoscope which is a long flexible narrow tube with a camera at the end is passed through the mouth, esophagus, stomach and the first part of the duodenum. The goal is to access a small elevation in the duodenum called the papilla of Vater. This papilla drains the biliary and pancreatic ducts which brings digestive juices from the liver, gallbladder and the pancreas. The endoscopist will inject contrast dye through the papilla into the ducts and takes X-rays to show lesions such as stones, strictures or blockages. If appropriate these can be treated by passing instruments through a port in the endoscope. Immediately following the endoscopic intervention; complications (bleeding, aspiration, perforation) will be recorded by study personnel as either yes or no, which will be used to assess the overall success of the procedure.

SUMMARY:
Post-ERCP pancreatitis is one of the most common complications accounting for substantial morbidity and mortality. The incidence of post-ERCP pancreatitis (PEP) has been studied in several large clinical trials and ranges from 1.6-15%. However most studies have demonstrated rates around 5%. This complication alone is estimated to cost the US healthcare around $150 million annually. To prevent this complication several pharmacological agents have been studied and no medication has been proved to be consistently effective in preventing this complications. Cyclo-oxygenase, and phospholipase A2 pathways are believed to play an important role in the pathogenesis of acute pancreatitis and so non-steroidal anti-inflammatory drugs (NSAIDs) have been extensively studied in the prevention of post-ERCP pancreatitis. One of the landmark studies done on prophylactic NSAIDs for PEP showed that rectal indomethacin significantly reduce the incidence of PEP (PEP developed in 9.2% vs. 16.9% of indomethacin and placebo groups respectively). Since then the use of rectal NSAIDs has become a standard chemo-prophylaxis for prevention of PEP especially in high risk patients. However, newly published meta-analysis showed that the role of peri-procedural rectal Indomethacin is doubtful in patients with average risk for PEP.

In this prospective randomized clinical study, we propose to study the effects of supplemental peri-operative oxygen on the incidence of PEP. The effects of high oxygen fraction (FIO2) has extensively been studied in reducing the incidence of surgical site infection, postoperative nausea, vomiting and to prevent postoperative atelectasis. Changing the FIO2 during a procedure can be a simple, inexpensive and low risk intervention to prevent post-procedure complications.

DETAILED DESCRIPTION:
The study will be a prospective, parallel-group, randomized double blinded control study conducted at University of Kentucky - Chandler Medical Center. Both the patient and the endoscopist will be blinded to the group assignment. Permuted block randomization will be used to randomly allocate a participant to a treatment group that will maintain a balance across treatment groups. Each block will have a specified number of randomly ordered treatment assignments. To assure randomization is blinded, randomization lists will be produced by the statistical team using varying block sizes of 100. Group assignments will be kept in sealed, sequentially numbered envelopes until used. Once patient is determined to be eligible, endoscopist will obtain consent and anesthetist will open the envelope which will assign patients either to Group 1: 30% FIO2 or Group 2: 80% FIO2. An anesthesia provider will administer FIO2 to the patient throughout the procedure period. Additional supplemental oxygen will be given to patients in either group at any time, as necessary, to maintain oxygen saturation as measured by pulse oximeter > 92%. Patients will be observed in the recovery area for at least 90 minutes after the procedure. Patients who develop abdominal pain during the post-endoscopy period are admitted to the hospital and standard pancreatitis clinical care is provided. Patients who are discharged after an uneventful ERCP will be contacted by telephone within 5 days to capture delayed occurrence of pancreatitis. Patients will again be contacted at 30 days to assess for delayed adverse events and to determine the severity of post-ERCP pancreatitis, which is defined in part by the length of hospitalization for pancreatitis.

Patients who do not consent to be included in the study will receive the standard endoscopic treatment at the discretion of the therapeutic endoscopist. The endoscopic intervention will be conducted in the endoscopy suite on the third floor at the University of Kentucky Healthcare medical center in Lexington, Kentucky. If no additional endoscopic intervention is required, then the patient will be scheduled for subsequent follow up clinic visits. After the conclusion of the study, patients will continue to be followed as clinically necessary by either the same or another gastroenterologist.

The patient has the right to withdraw consent to participate in the study at any time. The patient can be withdrawn from the study if they are not able to follow directions for study participation. If the patient decides to no longer take part in the study, their decision will have no effect on the medical care they will receive.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing ERCP
2. 18 years and older
3. capable of giving consent for the procedure

Exclusion Criteria:

1. Unwillingness or inability to consent for the study
2. Age less than 18 years
3. Standard contraindications to ERCP
4. Acute pancreatitis within 72hrs prior to ERCP
5. Chronic calcific pancreatitis
6. Pancreatic divisum
7. Pancreatic malignancy
8. ICU patients
9. Patients on home oxygen at baseline.
10. Incarcerated patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients with Post ERCP Pancreatitis | 2 months (90 minutes post-procedure to 2months follow-up)
  Patients will be observed in the recovery area for at least 90 minutes after the procedure. Patients who develop abdominal pain during the post-endoscopy period will be admitted to the hospital and standard pancreatitis clinical care is provided. Patients who are discharged after an uneventful ERCP will be contacted by telephone within 5 days to capture delayed occurrence of pancreatitis. Patients will again be contacted at 30 days to assess for delayed adverse events and to determine the severity of post-ERCP pancreatitis, which is defined in part by the length of hospitalization for pancreatitis. The patient participation in this study, which includes the endoscopy procedures and follow-up may last up to 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Moamen M. Gabr, MD, MSc, Principal Investigator — Assistant Professor, Internal Medicine, Gastroenterology
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loperfido S, Angelini G, Benedetti G, Chilovi F, Costan F, De Berardinis F, De Bernardin M, Ederle A, Fina P, Fratton A. Major early complications from diagnostic and therapeutic ERCP: a prospective multicenter study. Gastrointest Endosc. 1998 Jul;48(1):1-10. doi: 10.1016/s0016-5107(98)70121-x. PMID 9684657
- [Background] Masci E, Toti G, Mariani A, Curioni S, Lomazzi A, Dinelli M, Minoli G, Crosta C, Comin U, Fertitta A, Prada A, Passoni GR, Testoni PA. Complications of diagnostic and therapeutic ERCP: a prospective multicenter study. Am J Gastroenterol. 2001 Feb;96(2):417-23. doi: 10.1111/j.1572-0241.2001.03594.x. PMID 11232684
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Makela A, Kuusi T, Schroder T. Inhibition of serum phospholipase-A2 in acute pancreatitis by pharmacological agents in vitro. Scand J Clin Lab Invest. 1997 Aug;57(5):401-7. doi: 10.3109/00365519709084587. PMID 9279965
- [Background] Gross V, Leser HG, Heinisch A, Scholmerich J. Inflammatory mediators and cytokines--new aspects of the pathophysiology and assessment of severity of acute pancreatitis? Hepatogastroenterology. 1993 Dec;40(6):522-30. PMID 7509768
- [Background] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Background] Hovaguimian F, Lysakowski C, Elia N, Tramer MR. Effect of intraoperative high inspired oxygen fraction on surgical site infection, postoperative nausea and vomiting, and pulmonary function: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2013 Aug;119(2):303-16. doi: 10.1097/ALN.0b013e31829aaff4. PMID 23719611
- [Background] Testoni PA, Mariani A, Giussani A, Vailati C, Masci E, Macarri G, Ghezzo L, Familiari L, Giardullo N, Mutignani M, Lombardi G, Talamini G, Spadaccini A, Briglia R, Piazzi L; SEIFRED Group. Risk factors for post-ERCP pancreatitis in high- and low-volume centers and among expert and non-expert operators: a prospective multicenter study. Am J Gastroenterol. 2010 Aug;105(8):1753-61. doi: 10.1038/ajg.2010.136. Epub 2010 Apr 6. PMID 20372116
- See also: Major early complications from diagnostic and therapeutic ERCP: a prospective multicenter study. — https://www.ncbi.nlm.nih.gov/pubmed/9684657
- See also: Complications of diagnostic and therapeutic ERCP: a prospective multicenter study. — https://www.ncbi.nlm.nih.gov/pubmed/11232684
- See also: Incidence rates of post-ERCP complications: a systematic survey of prospective studies — https://www.ncbi.nlm.nih.gov/pubmed/17509029
- See also: Complications of endoscopic biliary sphincterotomy. — https://www.ncbi.nlm.nih.gov/pubmed/8782497
- See also: Inhibition of serum phospholipase-A2 in acute pancreatitis by pharmacological agents in vitro — https://www.ncbi.nlm.nih.gov/pubmed/9279965
- See also: Inflammatory mediators and cytokines--new aspects of the pathophysiology and assessment of severity of acute pancreatitis? — https://www.ncbi.nlm.nih.gov/pubmed/7509768
- See also: A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. — https://www.ncbi.nlm.nih.gov/pubmed/22494121
- See also: Effect of intraoperative high inspired oxygen fraction on surgical site infection, postoperative nausea and vomiting, and pulmonary function: systematic review and meta-analysis of randomized controlled trials. — https://www.ncbi.nlm.nih.gov/pubmed/23719611
- See also: Risk factors for post-ERCP pancreatitis in high- and low-volume centers and among expert and non-expert operators: a prospective multicenter study. — https://www.ncbi.nlm.nih.gov/pubmed/20372116